CLINICAL TRIAL: NCT00991081
Title: Exploratory/Developmental Study of Pharmacogenetic Smoking Cessation Therapy.
Brief Title: Behaviorally Enhanced Counseling on Nicotine Dependence (BEACON) Trial.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: SRI International (Industry); Johns Hopkins University (Other); University of Bristol (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-09152009-3940; 5R21DA027331-03 (NIH); Protocol # 16513 (Other: Stanford IRB)
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Results first posted 2012-09-19 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-08

CONDITIONS: Smoking
Keywords: pharmacogenetics; genetic counseling; genetic feedback; nicotine replacement; bupropion; smoking cessation; primary care; telehealth; motivational interviewing
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Counseling; Motivational Interviewing; Drug Therapy; Nicotine Replacement Therapy; Bupropion; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard treatment (Active Comparator): * Three 20-minute telephone calls during which a certified tobacco treatment specialist delivered motivationally-enhanced cognitive behavioral counseling.
  * A self-help guide for smoking cessation (Clearing the Air, NCI)sent by mail
  * A standard 8-week course of genetically-tailored pharmacotherapy
    * Participants with the A1 allele (TT/CT) were assigned to receive NRT (the Patch)
    * Participants with the A2 allele (CC) were assigned to receive bupropion
  Interventions: Behavioral: Counseling; Behavioral: Self-help guide; Drug: Pharmacotherapy
- Genetic feedback plus standard treatment (Experimental): In addition to the standard treatment, participants in this arm received the following interventions:
  * Genetic feedback, verbal - During the first counseling call, GF participants were informed of their genotype and provided with the rationale for their pharmacotherapy assignment
  * Genetic feedback, printed - After the first counseling call, GF participants were mailed a Personal Treatment Profile, which echoed each participant's ANNK1 genotype, the implications of this for smoking cessation treatment outcome, and which medication was chosen for them based on their genotype
  Interventions: Behavioral: Counseling; Behavioral: Self-help guide; Drug: Pharmacotherapy; Behavioral: Genetic feedback, verbal; Behavioral: Genetic feedback, printed

INTERVENTIONS:
Behavioral: Counseling — Three 20-minute telephone calls during which a certified tobacco treatment specialist delivered motivationally-enhanced cognitive behavioral counseling
  1. One week prior to the target quit date (TQD)
  2. Two weeks post-TQD
  3. Four weeks post-TQD
  Other Names: Motivational interviewing; Motivational enhancement
Behavioral: Self-help guide — A printed self-help guide for smoking cessation (Clearing the Air, NCI)sent by mail
  Other Names: Support Materials; Clearing the Air
Drug: Pharmacotherapy — 8-week course of genetically-tailored pharmacotherapy
  * Participants with the A1 allele (TT/CT) were assigned to receive NRT (the Patch)
  * Participants with the A2 allele (CC) were assigned to receive bupropion
  Other Names: NRT; Nicotine Replacement Therapy; The Patch; Bupropion; Zyban; Aplenzin; Wellbutrin
Behavioral: Genetic feedback, verbal — During the first counseling call, GF participants were informed of their genotype and provided with the rationale for their pharmacotherapy assignment
  Other Names: Pharmacogenetics; Pharmacogenetic counseling
  Arms: Genetic feedback plus standard treatment
Behavioral: Genetic feedback, printed — After the first counseling call, GF participants were mailed a Personal Treatment Profile, which echoed each participant's ANNK1 genotype, the implications of this for smoking cessation treatment outcome, and which medication was chosen for them based on their genotype.
  Other Names: Pharmacogenetics; Pharmacogenetic Feedback
  Arms: Genetic feedback plus standard treatment

SUMMARY:
The major purpose of this exploratory developmental study will be to develop a patient-centered and feasible protocol for communicating genetic data as it relates to drug efficacy for smoking cessation inpatients receiving medication that is matched to individual genotypes associated with increased efficacy for bupropion or nicotine replacement therapy.

DETAILED DESCRIPTION:
Therefore, our specific aims are to:

Aim 1: Conduct formative research to develop and refine a clinical protocol for a multi-component smoking cessation intervention, grounded in the extended parallel process model, consisting of pharmacogenetic treatment (smoking cessation drug matched to each individual smoker's genotype) and genetic feedback (delivery of patient-centered, personalized genotype information and its predictive value for smoking cessation treatment efficacy): We will adapt, pilot-test, and refine a theoretically-grounded PGx smoking cessation intervention using formative interviews of 20 African-American and European-ancestry smokers.

Aim 2: Conduct a mixed-methods feasibility trial randomizing treatment-seeking smokers to pharmacogenetic (PGx) treatment combined with genetic feedback (GF) vs. PGx treatment without GF for smoking cessation to examine the feasibility of the newly developed protocol in a primary care setting and characterize its psychological and behavioral impact: Smokers (N = 100) will be randomized to GF vs. no GF and all will receive motivational interviewing (standard care/SC) and PGx treatment. We will assess the impact of GF on time to relapse, medication adherence, and a comprehensive assessment battery of process and cognitive, psychological, and behavioral outcomes. Finally, we will synthesize quantitative and qualitative data to revise protocols, generate hypothesizes, and estimate effect sizes for a follow-up R01 submission.

ELIGIBILITY:
Inclusion and exclusion criteria are the same for participants in the formative interviews (Study A) and the feasibility RCT (Study B) except that Study A will include African American and European American smokers and Study B will include European American smokers.

Inclusion criteria:

* Adults (aged 18 or older)
* Currently smoke at least 10 cigarettes per day
* Motivated to quit smoking (>=5 on a 10-point Likert scale)
* Have a telephone
* Read and speak English.

Exclusion criteria:

* Any medical contraindications for transdermal nicotine replacement therapy (NRT) or sustained-release bupropion hydrochloride (bupropion) use based on the package labels (e.g., for bupropion, risk of seizure)
* DSM-IV Axis I diagnosis (other than nicotine dependence)
* Subjects who meet criteria for current major depression, or who demonstrate evidence of suicidal ideation at screening will be referred to treatment for depression and will be excluded from the study
* Must agree not to seek other treatment for smoking cessation during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean P David, MD SM DPhil, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - SRI International, Menlo Park, California
  - Stanford University School of Medicine, Stanford, California
  - Group Health Research Institute, Seattle, Washington

REFERENCES:
- [Result] McClure JB, Swan GE, St John J, Fauver R, Javitz HS, Bergen AW, Nishita D, Niaura R, Munafo MR, David SP. Pharmacogenetic smoking cessation intervention in a health care setting: a pilot feasibility study. Nicotine Tob Res. 2013 Feb;15(2):518-26. doi: 10.1093/ntr/nts173. Epub 2012 Sep 4. PMID 22949583

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase I and Phase II participants were recruited from members of Group Health Cooperative in Seattle, WA. Of the 36 Phase II participants enrolled, 32 had been previously genotyped for an earlier study and 4 were genotyped for this study.
Groups:
- Formative Interviews: Phase 1 involved formative research to develop and refine a patient-centered, theoretically grounded behavioral intervention for delivering genetically-tailored smoking cessation treatment. We convened a panel of doctorate level experts (n = 10) in pharmacogenetics; smoking cessation treatment; ethical, legal and social implications of genetics research; genetic literacy; patient-clinician communications; and mixed-methods research to guide development of the pharmacogenetic treatment, GF and evaluation.
  Next, smokers were asked about their familiarity with genetic concepts (e.g., DNA, genes), understanding of the roles genes play in smoking behavior and treatment response, reaction to the concept of genetically-tailoring pharmacotherapy, familiarity with the Genetic Information Nondiscrimination Act, concerns about privacy of genetic information, and interest in genetically-tailored treatment. Interviews were continued until response saturation was achieved (n = 10).
- Standard Treatment: Received behavioral counseling by telephone and either bupropion or nicotine replacement patch
- Genetic Feedback Plus Standard Treatment: Received genetic feedback regarding treatment selection in addition to behavioral counseling by telephone and either bupropion or nicotine replacement patch
Period: Phase I, Formative Research
Arm/Group | Formative Interviews | Standard Treatment | Genetic Feedback Plus Standard Treatment
Started | 20 | 0 | 0
Completed | 20 (The 10 smokers interviewed were not enrolled in the Phase II RCT.) | 0 | 0
Not Completed | 0 | 0 | 0
Period: Phase II, Randomized Control Trial
Arm/Group | Formative Interviews | Standard Treatment | Genetic Feedback Plus Standard Treatment
Started | 0 | 17 (Phase I interview participants were not enrolled in the Phase II RCT.) | 19 (Phase I interview participants were not enrolled in the Phase II RCT.)
Received First Clinical Call | 0 | 16 | 17
Completed | 0 | 15 | 15
Not Completed | 0 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment | Genetic Feedback Plus Standard Treatment | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 18 | 35
  >=65 years | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 49.4 (10.6) | 52.7 (8.22) | 51.1 (9.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Continuous Abstinence at 12 Weeks Post Target Quit Date
Description: Participants reporting continuous tobacco-use abstinence 12 weeks after their Target Quit Date, whose salivary cotinine levels confirmed their abstinence, were counted as "abstinent." All others were recorded as not abstinent.
Time Frame: 12 weeks after Target Quit Date
Population: All randomized participants were included in the data analysis.
Measure: Number; unit: participants
Groups:
- Standard Treatment: Received behavioral counseling by telephone, combined with either bupropion or nicotine replacement patch
- Genetic Feedback Plus Standard Treatment: Received genetic feedback regarding treatment selection in addition to behavioral counseling by telephone, combined with either bupropion or nicotine replacement patch
Arm/Group | Standard Treatment | Genetic Feedback Plus Standard Treatment
Number analyzed (Participants) | 17 | 19
participants | 3 | 2

2. Secondary Outcome: Morisky Adherence Scale
Description: Category: Treatment Acceptability Measures: Treatment Compliance Range: 0-8 Direction: Higher values represent higher compliance
Time Frame: 12 weeks after Target Quit Date
Population: Follow-up treatment satisfaction analyses includes only those participants not lost to follow-up (n = 30)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Treatment | Genetic Feedback Plus Standard Treatment
Number analyzed (Participants) | 15 | 15
units on a scale | 2.7 (1.9) | 1.8 (1.6)

3. Secondary Outcome: Trust Scale
Description: Category: Treatment Acceptability Measures: Trust in the clinician Range: 5-30 Direction: Higher values represent higher trust
Time Frame: Within 1 week of first clinical call
Population: First treatment satisfaction analyses include participants who received the first clinical call (n = 33)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Treatment | Genetic Feedback Plus Standard Treatment
Number analyzed (Participants) | 16 | 17
units on a scale | 19.3 (2.5) | 18.8 (2.3)

4. Secondary Outcome: Communication Scale
Description: Category: Treatment Acceptability Measures: Quality of verbal interaction and responsiveness during counseling sessions Range: 4-20 Direction: Higher values represent greater interaction and responsiveness
Time Frame: Within 1 week of first clinical call
Population: First treatment satisfaction analyses include participants who received the first clinical call (n = 33)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Treatment | Genetic Feedback Plus Standard Treatment
Number analyzed (Participants) | 16 | 17
units on a scale | 19.4 (1.4) | 19.4 (1.5)

5. Secondary Outcome: Satisfaction Scale
Description: Category: Treatment Acceptability Measures: Overall satisfaction with the clinician Range: 4-20 Direction: Higher values represent higher satisfaction
Time Frame: Within 1 week of first clinical call
Population: First treatment satisfaction analyses include participants who received the first clinical call (n = 33)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Treatment | Genetic Feedback Plus Standard Treatment
Number analyzed (Participants) | 16 | 17
units on a scale | 19.4 (1.8) | 19.5 (0.8)

6. Secondary Outcome: Treatment Interest Scale
Description: Category: Treatment Acceptability Measures: Interest in participating in recommended treatment plan Range: 1-10 Direction: Higher values represent higher treatment interest
Time Frame: Within 1 week of first clinical call
Population: First treatment satisfaction analyses include participants who received the first clinical call (n = 33)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Treatment | Genetic Feedback Plus Standard Treatment
Number analyzed (Participants) | 16 | 17
units on a scale | 9.0 (1.6) | 9.6 (0.74)

7. Secondary Outcome: Depression
Description: Category: Psychological Outcome Instrument: Center for Epidemiologic Studies Depression Scale (CES-D) Measures: Interest in participating in recommended treatment plan Range: 0-60 Direction: Higher values represent increased symptoms of depression
Time Frame: Within 1 week of first clinical call
Population: First psychological outcome analyses include participants who received the first clinical call (n = 30)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Treatment | Genetic Feedback Plus Standard Treatment
Number analyzed (Participants) | 16 | 17
units on a scale | 6.1 (7.8) | 4.1 (8.2)

8. Secondary Outcome: Fatalism
Description: Category: Psychological Outcome Instrument: Powe Fatalism Inventory, 10-item, revised Measures: belief in inevitability of smoking status Range: 0-10 Direction: Higher values represent increased fatalism beliefs
Time Frame: 12 weeks after Target Quit Date
Population: Follow-up psychological outcome analyses include only those participants not lost to follow-up (n = 30)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Treatment | Genetic Feedback Plus Standard Treatment
Number analyzed (Participants) | 15 | 15
units on a scale | 1.1 (1.8) | 0.4 (1.0)

9. Secondary Outcome: Intention to Quit
Description: Category: Psychological Outcome Instrument: 3-item inventory, Likert scale from 1 to 7 Measures: Intention, confidence, and expectation of quitting smoking Range: 3-21 Direction: Higher values represent increased intention to quit
Time Frame: Within 1 week of first clinical call
Population: First psychological outcome analyses include participants who received the first clinical call (n = 33)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Treatment | Genetic Feedback Plus Standard Treatment
Number analyzed (Participants) | 16 | 17
units on a scale | 18.3 (2.9) | 19.5 (1.9)

10. Secondary Outcome: Motivation
Description: Category: Psychological Outcome Instrument: Single item, Likert scale from 1 to 7 Measures: Desire to quit smoking Range: 1-7 Direction: Higher values represent increased motivation to quit
Time Frame: Within 1 week of first clinical call
Population: First psychological outcome analyses include participants who received the first clinical call (n = 33)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Treatment | Genetic Feedback Plus Standard Treatment
Number analyzed (Participants) | 16 | 17
units on a scale | 6.2 (1.0) | 6.4 (0.73)

11. Secondary Outcome: Perceived Control
Description: Category: Psychological Outcome Instrument: 3-item inventory, Likert scale from 1 to 7 Measures: Control over ability to quit smoking in the next month Range: 3-21 Direction: Higher values represent increased sense of control
Time Frame: Within 1 week of first clinical call
Population: First psychological outcome analyses include participants who received the first clinical call (n = 33)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Treatment | Genetic Feedback Plus Standard Treatment
Number analyzed (Participants) | 16 | 17
units on a scale | 14.0 (2.5) | 13.4 (3.4)

12. Secondary Outcome: Risk Perception
Description: Category: Psychological Outcome Instrument: 4-item inventory, Likert scale from 1 to 5 Measures: Perceived personal health risks from smoking Range: 4-20 Direction: Higher values represent increased perception of risk
Time Frame: Within 1 week of first clinical call
Population: First psychological outcome analyses include participants who received the first clinical call (n = 33)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Treatment | Genetic Feedback Plus Standard Treatment
Number analyzed (Participants) | 16 | 17
units on a scale | 15.3 (2.8) | 16.1 (2.5)

13. Secondary Outcome: Self-Efficacy
Description: Category: Psychological Outcome Instrument: 3-item inventory, Likert scale from 1 to 7 Measures: Perceived ability to quit smoking in the next month Range: 3-21 Direction: Higher values represent increased self-efficacy
Time Frame: Within 1 week of first clinical call
Population: First psychological outcome analyses include participants who received the first clinical call (n = 33)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Treatment | Genetic Feedback Plus Standard Treatment
Number analyzed (Participants) | 16 | 17
units on a scale | 16.2 (2.5) | 15.6 (2.6)

14. Secondary Outcome: Threat Minimization
Description: Category: Psychological Outcome Instrument: 2-item inventory, Likert scale from 1 to 7 Measures: Perceived presence of factors that would reduce personal smoking risks Range: 2-14 Direction: Higher values represent increased risk minimization
Time Frame: Within 1 week of first clinical call
Population: First psychological outcome analyses include participants who received the first clinical call (n = 33)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Treatment | Genetic Feedback Plus Standard Treatment
Number analyzed (Participants) | 16 | 17
units on a scale | 8.9 (2.9) | 7.3 (3.6)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Standard Treatment | Genetic Feedback Plus Standard Treatment
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 0/17 | 0/19

LIMITATIONS AND CAVEATS:
Possible selection bias as 32 of 36 participants had taken part in previous research

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No